CLINICAL TRIAL: NCT01395719
Title: Context - Remote Ischemic Conditioning in Renal Transplantation - Effect on Immediate and Extended Kidney Graft Function
Acronym: Context
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Sahlgrenska University Hospital (Other); Lundbeck Foundation (Other); Novo Nordisk A/S (Industry); AP Moeller Foundation (Other); Danish Society of Nephrology (Other); Aarhus University Hospital (Other); Erasmus Medical Center (Other); University Medical Center Groningen (Other); Danish Council for Independent Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 121369
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Transplantation; Delayed Graft Function; Acute Kidney Injury; Glomerular Filtration Rate
Keywords: renal transplantation; glomerular filtration rate; remote ischemic preconditioning; remote ischemic conditioning
MeSH Terms: conditions — Delayed Graft Function; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non remote ischemic conditionin(non-rIC) (No Intervention): Patients receiving kidney transplantation from a deceased donor. This group does not receive remote ischemic conditioning, but has a tourniquet on the leg (not inflated).
- Remote ischemic conditioning (rIC) (Experimental): Patients receiving kidney transplantation from a deceased donor. This group receives remote ischemic conditioning by inflating a tourniquet on the leg during surgery, before reperfusion of the kidney.
  Interventions: Other: Remote ischemic conditioning

INTERVENTIONS:
Other: Remote ischemic conditioning — Patients receiving kidney transplantation from a deceased donor. Remote ischemic conditioning (rIC) is done by inflating a tourniquet (250mmHg) on the patients leg before reperfusion of the kidney. The tourniquet stays on the leg on the opposite site of were the kidney is placed. rIC is done 4 x 5 min with 5 min intervals between with free blood flow.
  Other Names: Remote ischemic preconditioning; Ischemic conditioning
  Arms: Remote ischemic conditioning (rIC)

SUMMARY:
The purpose of this study is to determine whether remote ischemic conditioning can improve the outcome after renal transplantation with deceased donor. Remote ischemic conditioning is performed on the patient receiving a kidney from a deceased donor. Remote ischemic conditioning is done during the operation by inflating a tourniquet on the patients leg before opening the blood circulation to the kidney. The study focus on both the immediate kidney function after the transplantation, but also on the extended kidney function one year after the transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Received information, signed consent
* Candidate for kidney transplantation from deceased donor

Exclusion Criteria:

* Can't give informed consent
* AV-fistula in the leg opposite the site where the graft will be placed
* Threatening ischemia in the leg
* If donor is a small child
* If the patient receives a double transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Time to a 50% drop in baseline plasma-creatinine | minimum 1 week
  Plasma-creatinine changes posttransplant will be described using an exponential/logistic/linear model depending on the individual patient data. All plasma-creatinine values 30 days posttransplant, or in case of temporary posttransplant dialysis 30 days after the last performed dialysis, will be used, measured minimum twice daily initially. Baseline plasma-creatinine is measured approximately 1 hour prior to reperfusion of the kidney. Time to a 50% drop in baseline plasma-creatinine will be estimated.

SECONDARY OUTCOMES:
Need for dialysis | 1 week
GFR after 1 year | 12 months
  GFR measurement by Cr-EDTA.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoline V Krogstrup, MD, Principal Investigator — Klinisk Institut, Aarhus University; Bente Jespersen, Professor, DMSc, MD, Study Chair — Klinisk Institut, Aarhus University; Henrik Birn, DMSc, MD, Study Chair — University of Aarhus; Mihai Oltean, MD, PhD, Study Chair — Sahlgrenska University Hospital; Gertrude J. Nieuwenhuijs-Moeke, MD, Study Chair — University Medical Center Groningen; Frank J. M. F. Dor, MD, PhD, Study Chair — Erasmus Medical Center
Locations (4):
- Dept. of Renal Medicine, Aarhus University Hospital, Skejby, Aarhus N, Denmark
- Netherlands (2):
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Division of Transplant Surgery, Erasmus MC, University Medical Center, Rotterdam, Rotterdam
- Sahlgrenska Transplant Institute, Sahlgrenska Academy at the University of Gothenborg, Gothenburg, Sweden

REFERENCES:
- [Derived] Nielsen MB, Ravlo K, Eijken M, Krogstrup NV, Bue Svendsen M, Abdel-Halim C, Steen Petersen M, Birn H, Oltean M, Jespersen B, Moller BK. Dynamics of circulating dendritic cells and cytokines after kidney transplantation-No effect of remote ischaemic conditioning. Clin Exp Immunol. 2021 Nov;206(2):226-236. doi: 10.1111/cei.13658. Epub 2021 Sep 29. PMID 34473350
- [Derived] Nielsen MB, Jespersen B, Birn H, Krogstrup NV, Bourgonje AR, Leuvenink HGD, van Goor H, Norregaard R. Elevated plasma free thiols are associated with early and one-year graft function in renal transplant recipients. PLoS One. 2021 Aug 11;16(8):e0255930. doi: 10.1371/journal.pone.0255930. eCollection 2021. PMID 34379701
- [Derived] Nielsen MB, Krogstrup NV, Oltean M, Nieuwenhuijs-Moeke GJ, Dor FJMF, Birn H, Jespersen B. Remote ischaemic conditioning and early changes in plasma creatinine as markers of one year kidney graft function-A follow-up of the CONTEXT study. PLoS One. 2019 Dec 30;14(12):e0226882. doi: 10.1371/journal.pone.0226882. eCollection 2019. PMID 31887168
- [Derived] Nielsen MB, Krogstrup NV, Nieuwenhuijs-Moeke GJ, Oltean M, Dor FJMF, Jespersen B, Birn H. P-NGAL Day 1 predicts early but not one year graft function following deceased donor kidney transplantation - The CONTEXT study. PLoS One. 2019 Feb 28;14(2):e0212676. doi: 10.1371/journal.pone.0212676. eCollection 2019. PMID 30817778
- [Derived] Krogstrup NV, Oltean M, Nieuwenhuijs-Moeke GJ, Dor FJ, Moldrup U, Krag SP, Bibby BM, Birn H, Jespersen B. Remote Ischemic Conditioning on Recipients of Deceased Renal Transplants Does Not Improve Early Graft Function: A Multicenter Randomized, Controlled Clinical Trial. Am J Transplant. 2017 Apr;17(4):1042-1049. doi: 10.1111/ajt.14075. Epub 2016 Nov 9. PMID 27696662
- [Derived] Krogstrup NV, Oltean M, Bibby BM, Nieuwenhuijs-Moeke GJ, Dor FJ, Birn H, Jespersen B. Remote ischaemic conditioning on recipients of deceased renal transplants, effect on immediate and extended kidney graft function: a multicentre, randomised controlled trial protocol (CONTEXT). BMJ Open. 2015 Aug 20;5(8):e007941. doi: 10.1136/bmjopen-2015-007941. PMID 26297360